CLINICAL TRIAL: NCT05681000
Title: Phase I Clinical Study on the Tolerability of Utidelone Capsule in Patients With Advanced Solid Tumors
Brief Title: Tolerability of Utidelone Capsule in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biostar Pharma, Inc. (Industry)
Responsible Party: Sponsor
Organization: Beijing Biostar Pharmaceuticals Co., Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG02-2201
Record Dates: First submitted 2022-12-30; First posted 2023-01-11 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: At least 4 dose cohorts are planned, and 16-28 cases are expected.
  1. Cohort 1: 2 subjects are planned to take 25 mg/m2/d by QD for 5 consecutive days in a 21-day cycle.
  2. Cohort 2: 2 subjects are planned to take 50 mg/m2/d by QD for 5 consecutive days in a 21-day cycle.
  3. Cohort 3: 3-6 subjects are planned to take 75 mg/m2/d by QD for 5 consecutive days in a 21-day cycle.
  4. Cohort 4: 3-6 subjects are planned to take 100 mg/m2/d by QD for 5 consecutive days in a 21-day cycle.
  5. Cohort 5: 3-6 subjects are planned to take 100 mg/m2/d by QD for 7 consecutive days in a 21-day cycle.
  6. Cohort 6: 3-6 subjects are planned to take 120 mg/m2/d by QD for 7 consecutive days in a 21-day cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Utidelone Capsule at 25 mg/m2/d for 5 days (Experimental): Cohort 1: 2 subjects are planned to take Utidelone Capsule at 25 mg/m2/d by QD for 5 consecutive days in a 21-day cycle.
  Interventions: Drug: Utidelone Capsule
- Utidelone Capsule at 50 mg/m2/d for 5 days (Experimental): Cohort 2: 2 subjects are planned to take Utidelone Capsule at 50 mg/m2/d by QD for 5 consecutive days in a 21-day cycle.
  Interventions: Drug: Utidelone Capsule
- Utidelone Capsule at 75 mg/m2/d for 5 days (Experimental): Cohort 3: 3-6 subjects are planned to take Utidelone Capsule at 75 mg/m2/d by QD for 5 consecutive days in a 21-day cycle.
  Interventions: Drug: Utidelone Capsule
- Utidelone Capsule at 100 mg/m2/d for 5 days (Experimental): Cohort 4: 3-6 subjects are planned to take Utidelone Capsule at 100 mg/m2/d by QD for 5 consecutive days in a 21-day cycle.
  Interventions: Drug: Utidelone Capsule
- Utidelone Capsule at 100 mg/m2/d for 7 days (Experimental): Cohort 5: 3-6 subjects are planned to take Utidelone Capsule at 100 mg/m2/d by QD for 7 consecutive days in a 21-day cycle.
  Interventions: Drug: Utidelone Capsule
- Utidelone Capsule at 120 mg/m2/d for 7 days (Experimental): Cohort 6: 3-6 subjects are planned to take Utidelone Capsule at 120 mg/m2/d by QD for 7 consecutive days in a 21-day cycle.
  Interventions: Drug: Utidelone Capsule

INTERVENTIONS:
Drug: Utidelone Capsule — At least 4 dose cohorts are planned, and 16-28 cases are expected.
  1. Cohort 1 and 2: 2 cases are planned for each. In cohort 1, the subjects will receive Utidelone Capsule at a dose of 25 mg/m2/d for 5 days, in a 21-day cycle. In cohort 2, the subjects will receive Utidelone Capsule at a dose of 50 mg/m2/d for 5 days, in a 21-day cycle.
  2. Other dose-escalation cohorts: 3-6 cases are planned in each cohort, following the 3 + 3 design. The subjects in these cohorts will receive Utidelone Capsule at 75 mg/m2/d for 5 days, 100 mg/m2/d for 5 days, 100 mg/m2/d for 7 days, and 120 mg/m2/d for 7 days in a 21-day cycle respectively.

SUMMARY:
The purpose of this trial is to evaluate the safety and tolerability of Utidelone Capsule in patients with advanced solid tumors and determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT). The secondary objectives are to evaluate the pharmacokinetic profile of Utidelone Capsule in patients with advanced solid tumors, preliminarily assess the anti-tumor activity of Utidelone Capsule in patients with advanced solid tumors via objective radiologic tumor response using RECIST 1.1, and to recommend the dose and dosage regimen for subsequent clinical trials.

DETAILED DESCRIPTION:
At least 4 dose cohorts are planned, and 16-28 cases are expected.

1. Cohort 1 and 2: 2 cases are planned for each.
2. Other dose-escalation cohorts: 3-6 cases are planned in each cohort, following the 3 + 3 design.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to sign a written informed consent;
2. Patients with histologic or pathologic documentation of incurable, locally advanced, or metastatic solid tumors for which standard therapies are not available, no longer effective, and not tolerated, and for those patients who have declined the standard therapies;
3. Male or female subjects aged ≥18, with ECOG performance status scored 0-1;
4. Expected survival time ≥ 12 weeks;
5. Adequate organ and marrow function as defined below:

   1. neutrophil count (ANC) ≥ 1.5 × 109/L
   2. platelet count (PLT) ≥ 100 × 109/L
   3. hemoglobin ≥ 9 g/dL
   4. total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN)
   5. alanine transaminase (ALT) ≤ 2.5 × ULN
   6. aspartate transaminase (AST) ≤ 2.5 × ULN
   7. Creatinine clearance ≥ 60 mL/min
6. Female patients of childbearing potential must have negative serum or urine pregnancy test at screening;
7. Sexually active women, unless surgically sterile (at least 6 months prior to study drug administration) or postmenopausal for at least 12 consecutive months, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives [any hormonal method in conjunction with a secondary method], intrauterine device, female condom with spermicide, diaphragm with spermicide, absolute sexual abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to Study drug administration] sexual partner) for at least 4 weeks prior to study drug administration, during study and up to 30 days or till next chemotherapy cycle. Cessation of birth control after this point should be discussed with a responsible physician. Investigator will discuss with patient on the above points and the patient agreement will be documented in the source document. The investigator should ensure that the patient is using an effective method of avoiding pregnancy as per protocol. In case of Male patients: Either patient partners or patients themselves must use an effective method of avoiding pregnancy for at least 4 weeks prior to study drug administration, during study and up to 30 days or till next chemotherapy cycle.

Exclusion Criteria:

1. Patients who have received non-investigational anti-tumor therapies (such as chemotherapy, radiotherapy, immunotherapy, biological therapy or traditional Chinese medicine treatment) within 2 weeks prior to study drug administration;
2. Patients with hypersensitivity reaction caused by previous anti-microtubule drugs;
3. Patients who have known brain metastasis; patients whose CNS metastases have been treated by surgery or radiotherapy, who are no longer on corticosteroids, and who are neurologically stable are eligible;
4. Patients with a history of the following within 6 months prior to Cycle 1 Day 1: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) Class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or ECG abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder. Atrial fibrillation is allowed if rate is controlled;
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements;
6. Patients with baseline QTc interval > 470 msec;
7. Patients with known history of human immunodeficiency virus (HIV) infection with an exception that if they have not had an opportunistic infection within the past 12 months, they are eligible;
8. Patients who are HBV DNA positive;
9. Patients with pre-existing > Grade 1 peripheral sensory neuropathy (NCI CTCAE 5.0) ;
10. Patients who still experience ≥ Grade 2 acute toxicities caused by previous anti-tumor therapies (e.g. chemotherapy, radiotherapy, immunotherapy, biological therapy or TCM treatment) prior to enrollment (NCI-CTCAE 5.0, except alopecia);
11. Patients who have undergone any major surgery or have major trauma within 4 weeks prior to administration of the investigational product or are expected to undergo major surgery during the first cycle of treatment;
12. Patients who have received other investigational treatments within 4 weeks prior to administration of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose, MTD | 12 months
  The maximum tolerated dose (MTD) is defined as the highest dose tested in which none or only one patient experienced DLT attributable to the study drug(s), when 6 patients were treated at that dose and are evaluable for toxicity. The MTD is one dose level below the lowest dose tested in which 2 or more patients experienced DLT attributable to the study drug(s).
Dose-Limiting Toxicity, DLT | 12 months
  DLT is observed during Cycle 1 in the dose escalation trial. Any toxicity meeting the criteria outlined in the protocol, at least possibly related to study drug (i.e. definitely, probably, or possibly attributed), will be considered a DLT.

SECONDARY OUTCOMES:
Maximum (or peak) serum concentration-Cmax | 12 months
  Cmax of Utidelone Capsule
Time to peak drug concentration-Tmax | 12 months
  Tmax of Utidelone Capsule
the area under the concentration-time curve from dosing (time 0) to time t-AUC0-t | 12 months
  the AUC0-t of Utidelone Capsule
the time required for plasma concentration of a drug to decrease by 50%-t1/2 | 12 months
  the t1/2 of Utidelone Capsule
Objective Response Rate-ORR | 12 months
  The percentage of patients who have a partial response or complete response to the treatment within a certain period of time.
Recommended Phase II Dose (RP2D) | 12 months
  To recommend the dose and dose regimen for subsequent clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Thomas, MD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States